CLINICAL TRIAL: NCT05647304
Title: Pilot Clinical Investigation Evaluating the Safety and Performance of RGn550 in Treating Sportspeople Suffering From Acute Concussion Syndrome - A Prospective, Comparative, Randomized, Simple-blinded, Monocentric Investigation [RGncon Investigation]
Brief Title: Pilot Clinical Investigation Evaluating the Safety and Performance of RGn550 in Treating Sportspeople Suffering From Acute Concussion Syndrome
Acronym: RECOVERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: REGEnLIFE SAS (Industry)
Collaborators: RCTs (Industry); University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RGnCON; 2022-A01319-34 (Registry Identifier: IDRCB number. French competent authority : Agence Nationale de sécurité du médicament et des produits de santé (ANSM))
Record Dates: First submitted 2022-11-22; First posted 2022-12-12 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-10

CONDITIONS: Acute Concussion Syndrome
Keywords: Concussion; mTBI; Neurostimulation; Optics and photonics; Photobiomodulation; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Medical Device
MeSH Terms: conditions — Brain Concussion; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: An interventional, prospective, monocentric, randomized, comparative and simple-blinded pilot clinical investigation
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 Hz-PWM (Other): RGn550 with a 5 Hz-pulsed wave mode light emission
  Interventions: Device: RGn550 5 Hz-PWM
- 10 Hz-PWM (Other): RGn550 with a 10 Hz-pulsed wave mode light emission
  Interventions: Device: RGn550 10 Hz-PWM

INTERVENTIONS:
Device: RGn550 5 Hz-PWM — RGn550 with a 5 Hz-pulsed wave mode light emission
  Arms: 5 Hz-PWM
Device: RGn550 10 Hz-PWM — RGn550 with a 10 Hz-pulsed wave mode light emission
  Arms: 10 Hz-PWM

SUMMARY:
This is a controlled investigation, with randomization of the patients, which aims at evaluating the safety and performance of device RGn550 in treating sportspeople suffering from acute concussion syndrome. RGn550 is a non-invasive medical device which is applied on the head (helmet). It combines 2 technologies:

* PhotoBioModulation (PBM), which involves exposure to light from the red to near-infrared wavelengths using lasers and Light Emitting Diodes (LEDs)
* Static Magnetic Stimulation (SMS), which consists in the application of a static magnetic field.

Considering previous investigations, this innovative technology could reduce brain inflammation implicated in concussion syndrome.

DETAILED DESCRIPTION:
This monocentric investigation is planned to include 50 patients who will be followed up to 52 days.

Patients meeting all eligibility criteria will be randomized on a 1: 1 ratio into one of the two groups differing in terms of light exposure duty cycle (duty cycle is 50%) treatment frequency: RGn550 device with a 5 Hz-pulsed wave mode light emission frequency and RGn550 device with a 10 Hz-pulsed wave mode light emission frequency. The RGn550 device will be applied to the patients during two 20-min treatment sessions at 1 week apart.

Three onsite visits will be performed at the following timepoints:

* Day 0 (D0): Inclusion, randomization (to the 5 Hz-PWM or 10Hz-PWM treatment group) and first treatment session with RGn550
* Day 7 (D7): Second treatment session with RGn550
* Day 52 (D52): Evaluation 45 days after the last treatment session. In addition, at Day 14 (D14), the patient will be asked to remotely assess his/her concussion syndrome symptoms.

At inclusion visit, after verification of the eligibility criteria, data regarding patients will be collected: demographic data, result of pregnancy test for women, concussion history, concomitant medications.

At each visit:

* The patient will be asked to assess his/her concussion syndrome symptoms via the SCAT5 evaluation tool
* The functions possibly affected by the concussion syndrome will be assessed at each visit:

O The executive function via the TMT A&B O The automated oculomotor and oculopostural functions via the NPC, cover test and Maddox Rod test O The balance via static stabilometric tests

•all AEs and device deficiencies will be collected A blood sample will be collected at D0 and D52 to measure blood markers of concussion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged at least 18 years old
* Suffering from concussion syndrome resulting from a shock that occurred during sport practice less than 72h ago, as confirmed by neurological examination via the Head Injury Assessment - Form 3 (HIA3) tool
* Affiliated to French social security
* Who provided a dated and signed informed consent form.

Non-inclusion Criteria:

* Patient protected by a French legal measure ("sauvegarde de justice", "tutelle" or "curatelle")
* Patient not able to express his/her consent
* Patient deprived of liberty or hospitalized without consent
* Woman who is pregnant or breastfeeding, or who plans to become pregnant or breastfeeding during the investigation, or who has the capacity to conceive but is not using a reliable contraceptive method as deemed by the investigator
* Patient living in a medical facility
* Patient who experienced a surgery at the treatment application area (head) within 3 months prior to inclusion
* Patient with skin lesions on the treatment application area (head)
* Patient with a short-term life-threatening pathology (e.g., evolving cancer; non-stable heart failure; severe hepatic, renal or respiratory failure, etc.)
* Patient diagnosed with a heart attack within 3 months prior to inclusion
* Patient implanted with ferromagnetic material
* Patient implanted with a pacemaker
* Patient with a risk of epileptic seizure or other non-degenerative central nervous system diseases
* Patient with major physical or neurosensorial disorders that may interfere with assessments
* Patient with chronic psychosis or psychotic episodes
* Patient addicted to alcohol or drugs
* Patient treated with antidepressant or benzodiazepine
* Patient who participated to another investigation/study involving the use of an investigational medical device/drug within the 30 days prior inclusion
* Patient not able to meet treatment sessions as deemed by the investigator
* Patient not able to complete requested investigation assessments as deemed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period : 11 October 2022 - 02 May 2023 One site located in France
Period: Overall Study
Arm/Group | 5 Hz-PWM | 10 Hz-PWM
Started | 26 | 24
Completed | 25 | 24
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients randomized and treated at least once (at the inclusion visit)
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 Hz-PWM | 10 Hz-PWM | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (5.2) | 25.1 (5.1) | 25.0 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 23 | 21 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 26 | 24 | 50
Time between concussion and inclusion [Mean (Standard Deviation); unit: days] | 2.4 (0.5) | 2.3 (0.4) | 2.3 (0.5)
Concussion history [Mean (Standard Deviation); unit: concussion] | 2.0 (2.1) | 1.4 (1.6) | 1.7 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of RGn550's Adverse Device Effects (ADEs)
Description: Percentage of patients with at least one ADE
Time Frame: Throughout the investigation (from Day 0 to Day 52)
Population: Patients randomized and treated at least once (at inclusion visit)
Measure: Count of Participants; unit: Participants
Arm/Group | 5 Hz-PWM | 10 Hz-PWM
Number analyzed (Participants) | 26 | 24
Participants | 10 | 10

2. Secondary Outcome: Incidence of RGn550's ADEs Per Severity (Mild, Moderate and Severe)
Description: Percentage of patients with at least one ADE per severity (mild, moderate and severe)
Time Frame: Throughout the investigation (from Day 0 to Day 52)
Population: Patients randomized and treated at least once (at inclusion visit)
Measure: Count of Participants; unit: Participants
Arm/Group | 5 Hz-PWM | 10 Hz-PWM
Number analyzed (Participants) | 26 | 24
Participants
  Patients who had at least one mild ADE | 10 | 10
  Patients who had at least one moderate ADE | 0 | 0
  Patients who had at least one severe ADE | 0 | 0

3. Secondary Outcome: Incidence of RGn550's Adverse Events (AEs)
Description: Percentage of patients with at least one AE
Time Frame: Throughout the investigation (from Day 0 to Day 52)
Population: Patients randomized and treated at least once (at inclusion visit)
Measure: Count of Participants; unit: Participants
Arm/Group | 5 Hz-PWM | 10 Hz-PWM
Number analyzed (Participants) | 26 | 24
Participants | 12 | 10

4. Secondary Outcome: Incidence of RGn550's Device Deficiencies (DDs)
Description: Percentage of patients with at least one DD
Time Frame: Throughout the investigation (from Day 0 to Day 52)
Population: Patients randomized and treated at least once (at inclusion visit)
Measure: Count of Participants; unit: Participants
Arm/Group | 5 Hz-PWM | 10 Hz-PWM
Number analyzed (Participants) | 26 | 24
Participants | 4 | 1

5. Secondary Outcome: Evolution of Automated Oculomotor and Oculopostural Functions, as Assessed Through the Convergence
Description: Evolution of the Near Point of Convergence (NPC)
Time Frame: at Day 0 and Day 7 (before and after treatment session) and at Day 52
Population: Patients randomized and treated at least once (at inclusion visit)
Measure: Mean (Standard Deviation); unit: NPC (cm)
Arm/Group | 5 Hz-PWM | 10 Hz-PWM
Number analyzed (Participants) | 26 | 24
NPC (cm)
  D0 before treatment | 4.6 (5.6) | 2.9 (3.1)
  D0 after treatment | 1.8 (2.6) | 0.4 (1.2)
  D7 before treatment: number analyzed (Participants) | 25 | 24
  D7 before treatment | 1.3 (2.1) | 0.3 (0.8)
  D7 after treatment: number analyzed (Participants) | 25 | 24
  D7 after treatment | 1.0 (1.8) | 0.1 (0.4)
  D52: number analyzed (Participants) | 25 | 24
  D52 | 0.9 (1.8) | 0.4 (1.0)

6. Secondary Outcome: Evolution of Automated Oculomotor and Oculopostural Functions, as Assessed Through Deviations
Description: Evolution of the deviation assessed via the Cover test considering both eyes
  The unilateral cover test was used in this investigation, which consists into covering one eye, horizontally moving a target 5 cm in front of both eyes, and then uncovering the covered eye and observing its reaction. If it fixes the target, this is normal: there is an orthophoria. If it moves to fix the target (restitution movement), the test is positive: there is a heterophoria in near vision. Patients who had visual corrections were to keep them during the test. The test was then repeated on the other eye.
  The outcome of this test was a deviation value, considering both eyes, comprised between 0 (better outcome = normal fixation) and 3 (worst outcome = deviated eye without restitution movement).
Time Frame: at Day 0 and Day 7 (before and after treatment session) and at Day 52
Population: Patients randomized and treated at least once (at inclusion visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5 Hz-PWM | 10 Hz-PWM
Number analyzed (Participants) | 26 | 24
score on a scale
  D0 before treatment | 1.5 (0.9) | 1.5 (1.0)
  D0 after treatment | 0.9 (1.0) | 1.0 (1.0)
  D7 before treatment: number analyzed (Participants) | 25 | 24
  D7 before treatment | 1.0 (0.9) | 0.8 (1.0)
  D7 after treatment: number analyzed (Participants) | 25 | 24
  D7 after treatment | 0.6 (1.0) | 0.6 (0.8)
  D52: number analyzed (Participants) | 25 | 24
  D52 | 0.8 (1.1) | 0.5 (0.8)

7. Secondary Outcome: Evolution of Automated Oculomotor and Oculopostural Functions, as Assessed Through Deviations
Description: Evolution of the deviations assessed via Maddox rod test (horizontal deviation, vertical deviation of at least one eye)
Time Frame: at Day 0 and Day 7 (before and after treatment session) and at Day 52
Population: Patients randomized and treated at least once (at inclusion visit)
Measure: Count of Participants; unit: Participants
Arm/Group | 5 Hz-PWM | 10 Hz-PWM
Number analyzed (Participants) | 26 | 24
Participants
  Horizontal deviation : D0 before treatment | 18 | 17
  Horizontal deviation : D0 after treatment | 11 | 13
  Horizontal deviation : D7 before treatment: number analyzed (Participants) | 25 | 24
  Horizontal deviation : D7 before treatment | 12 | 11
  Horizontal deviation : D7 after treatment: number analyzed (Participants) | 25 | 24
  Horizontal deviation : D7 after treatment | 10 | 10
  Horizontal deviation : D52: number analyzed (Participants) | 25 | 24
  Horizontal deviation : D52 | 11 | 14
  Vertical deviation of at least one eye : D0 before treatment | 9 | 7
  Vertical deviation of at least one eye : D0 after treatment | 4 | 4
  Vertical deviation of at least one eye : D7 before treatment: number analyzed (Participants) | 25 | 24
  Vertical deviation of at least one eye : D7 before treatment | 4 | 1
  Vertical deviation of at least one eye : D7 after treatment: number analyzed (Participants) | 25 | 24
  Vertical deviation of at least one eye : D7 after treatment | 2 | 1
  Vertical deviation of at least one eye : D52: number analyzed (Participants) | 25 | 24
  Vertical deviation of at least one eye : D52 | 3 | 1

8. Secondary Outcome: Evolution of the Balance Function, as Assessed Through Static Stabilometric Parameters
Description: Evolution of statokinesigram area with closed eyes
  The statokinesigram is the projection onto a 2-dimensional space of the trajectory of the patient's center of pressure. Its area is measured in mm2. The larger the area is, the higher the patient's imbalance is.
  The statokinesigram area was measured using the stabilometric platform KFORCE Plates on which the patients were asked to stand for 30 s with closed eyes.
Time Frame: at Day 0 and Day 7 (before and after treatment session) and at Day 52
Population: Patients randomized and treated at least once (at inclusion visit)
Measure: Mean (Standard Deviation); unit: mm2
Arm/Group | 5 Hz-PWM | 10 Hz-PWM
Number analyzed (Participants) | 25 | 24
mm2
  D0 before treatment | 51.9 (28.9) | 54.9 (41.4)
  D0 after treatment | 64.4 (50.5) | 62.9 (60.2)
  D7 before treatment: number analyzed (Participants) | 24 | 24
  D7 before treatment | 51.0 (34.3) | 56.8 (33.2)
  D7 after treatment: number analyzed (Participants) | 24 | 24
  D7 after treatment | 47.9 (31.2) | 59.9 (41.9)
  D52: number analyzed (Participants) | 24 | 24
  D52 | 50.9 (33.9) | 51.9 (39.5)

9. Secondary Outcome: Evolution of the Balance Function, as Assessed Through Static Stabilometric Parameters
Description: Evolution of the difference between left and right distributions of patient's body weight
  Patient's body weight left distribution, respectively right distribution, refer to patient's body weight distribution on his/her left foot, respectively right foot.
  The left distribution and the right distribution are two percentages which sum makes 100%.
  When body weight is well distributed between left and right feet (coherent balance), the difference between left and right distributions is ≤ 5%.
  When body weight is not well distributed between left and right feet (uncoherent balance), the difference between left and right distributions is > 5%.
  These distributions were measured using the stabilometric platform KFORCE Plates on which the patients were asked to stand for 30 s with closed eyes.
Time Frame: at Day 0 and Day 7 (before and after treatment session) and at Day 52
Population: Patients randomized and treated at least once (at inclusion visit)
Measure: Mean (Standard Deviation); unit: % of body weight distribution difference
Arm/Group | 5 Hz-PWM | 10 Hz-PWM
Number analyzed (Participants) | 26 | 24
% of body weight distribution difference
  D0 before treatment | 6.5 (4.1) | 6.3 (4.7)
  D0 after treatment | 6.9 (4.3) | 6.3 (5.0)
  D7 before treatment: number analyzed (Participants) | 25 | 24
  D7 before treatment | 5.7 (3.5) | 7.5 (5.7)
  D7 after treatment: number analyzed (Participants) | 25 | 24
  D7 after treatment | 5.0 (4.7) | 5.2 (4.1)
  D52: number analyzed (Participants) | 25 | 24
  D52 | 6.0 (5.1) | 6.4 (4.5)

10. Secondary Outcome: Evolution of Executive Function, as Assessed With the Trail Making Test Part A and B (TMT A&B)
Description: Evolution of the Trail Making Test part A and B (TMT A&B) time to perform the task
Time Frame: at Day 0 (before treatment session) and at Day 7 (after treatment session) Of note: for 46 patients, TMTB was performed before (rather than after) treatment at D7 (deviation)
Population: Patients randomized and treated at least once (at inclusion visit)
Measure: Mean (Standard Deviation); unit: s
Arm/Group | 5 Hz-PWM | 10 Hz-PWM
Number analyzed (Participants) | 26 | 24
s
  TMTA time to perform the task: D0 | 19.0 (5.4) | 21.2 (7.0)
  TMTA time to perform the task: D7: number analyzed (Participants) | 25 | 24
  TMTA time to perform the task: D7 | 15.7 (4.0) | 18.5 (4.8)
  TMTB time to perform the task: D0 | 53.5 (20.1) | 50.9 (26.6)
  TMTB time to perform the task: D7: number analyzed (Participants) | 25 | 24
  TMTB time to perform the task: D7 | 42.5 (12.7) | 43.1 (17.9)

11. Secondary Outcome: Evolution of Concussion Syndrome Symptoms
Description: Evolution of the SCAT5 (Sport Concussion Assessment Tool - 5th edition) score
  The SCAT5 is a standardized tool for evaluating concussions designed for use by physicians and licensed healthcare professionals. With this tool, the patient rates the intensity of every symptom from 0 (none) to 6 (severe) using a form. This enables to calculate the total number of symptoms (subscore from 0 to 22) and the symptom severity score (subscore from 0 to 132).
Time Frame: at baseline (which represents the patient's state before the concussion as estimated/assessed by the patient on D0), Day 0 (before treatment session), Day 7 (before treatment session), Day 14 and Day 52
Population: Patients randomized and treated at least once (at inclusion visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5 Hz-PWM | 10 Hz-PWM
Number analyzed (Participants) | 26 | 24
score on a scale
  Total number of symptoms: baseline | 0.4 (0.8) | 0.3 (0.4)
  Total number of symptoms : D0 before treatment | 4.6 (3.7) | 5.5 (4.7)
  Total number of symptoms : D7 before treatment: number analyzed (Participants) | 25 | 24
  Total number of symptoms : D7 before treatment | 1.2 (2.2) | 1.7 (4.2)
  Total number of symptoms : D14: number analyzed (Participants) | 25 | 24
  Total number of symptoms : D14 | 0.4 (1.1) | 1.3 (4.0)
  Total number of symptoms : D52: number analyzed (Participants) | 25 | 24
  Total number of symptoms : D52 | 0.2 (0.6) | 0.8 (3.1)
  Symptom severity score: baseline | 0.7 (1.5) | 0.4 (0.8)
  Symptom severity score: D0 before treatment | 7.5 (7.4) | 10.8 (13.2)
  Symptom severity score: D7 before treatment: number analyzed (Participants) | 25 | 24
  Symptom severity score: D7 before treatment | 2.1 (4.2) | 3.5 (11.9)
  Symptom severity score: D14: number analyzed (Participants) | 25 | 24
  Symptom severity score: D14 | 0.8 (2.2) | 2.9 (11.1)
  Symptom severity score: D52: number analyzed (Participants) | 25 | 24
  Symptom severity score: D52 | 0.3 (1.2) | 2.1 (9.2)

12. Secondary Outcome: Evolution of the Concussion Blood Markers
Description: Evolution of the concentration of:
  * Anti-inflammatory cytokines InterLeukin (IL)-1 receptor antagonist, IL-4, IL-6, IL-10, IL-11 and IL-13
  * S100 calcium binding protein B (S100B)
  * Glial Fibrillary Acidic Protein (GFAP)
  * Ubiquitin C-terminal Hydrolase-L1 (UCH-L1) Of note: IL-11 and IL-13 could eventually not be analyzed due to undetectable low concentrations
Time Frame: at Day 0 (before treatment session) and at Day 52
Population: Patients randomized and treated at least once (at inclusion visit)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | 5 Hz-PWM | 10 Hz-PWM
Number analyzed (Participants) | 26 | 24
pg/mL
  GFAP : D0 before treatment | 95.3 (75.6) | 82.5 (40.2)
  GFAP : D52: number analyzed (Participants) | 25 | 24
  GFAP : D52 | 67.7 (29.6) | 49.8 (21.5)
  UCHL1 : D0 before treatment | 11.0 (20.4) | 3.9 (4.4)
  UCHL1 : D52: number analyzed (Participants) | 25 | 24
  UCHL1 : D52 | 9.3 (13.3) | 5.0 (4.5)
  IL-1RA : D0 before treatment | 367.8 (231.8) | 413.3 (318.7)
  IL-1RA : D52: number analyzed (Participants) | 25 | 24
  IL-1RA : D52 | 324.2 (122.5) | 452.5 (423.8)
  IL-10 : D0 before treatment | 0.74 (1.88) | 0.33 (0.16)
  IL-10 : D52: number analyzed (Participants) | 25 | 24
  IL-10 : D52 | 0.28 (0.08) | 0.51 (0.47)
  IL-4 : D0 before treatment | 0.02 (0.01) | 0.02 (0.01)
  IL-4 : D52: number analyzed (Participants) | 25 | 24
  IL-4 : D52 | 0.05 (0.05) | 0.05 (0.04)
  IL-6 : D0 before treatment: number analyzed (Participants) | 25 | 24
  IL-6 : D0 before treatment | 1.25 (2.32) | 2.36 (3.44)
  IL-6 : D52: number analyzed (Participants) | 25 | 24
  IL-6 : D52 | 0.97 (1.85) | 1.35 (2.19)
  S100B : D0 before treatment | 25.7 (35.4) | 17.6 (10.9)
  S100B : D52: number analyzed (Participants) | 25 | 24
  S100B : D52 | 25.0 (36.0) | 17.2 (10.5)

ADVERSE EVENTS:
Time Frame: Throughout the investigation (from D0 to D52)
Arm/Group | 5 Hz-PWM | 10 Hz-PWM
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 12/26 | 10/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 Hz-PWM (N=26) | 10 Hz-PWM (N=24)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Medical device site discomfort (General disorders) | 5 (5) | 4 (4)
Medical device site warmth (General disorders) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 6 (6) | 8 (9)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Lack of sham group Single blinding Monocentric design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the investigators wish to publish data from this investigation (poster, abstract, article, etc.), they must first seek approval from REGEnLIFE.

DOCUMENTS (2):
  • Study Protocol (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT05647304/Prot_002.pdf
  • Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT05647304/SAP_003.pdf